CLINICAL TRIAL: NCT04035980
Title: Clinical Trial to Evaluate Efficacy and Acceptance of a Telemedicine Based Programme to Treat Hepatitis C Among Patients at Drug Addiction Centers
Brief Title: Telemedicine for Linkage to Care People Who Injected Drugs With Hepatitis C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, Principal Investigator, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telemedicine_HCV
Record Dates: First submitted 2019-07-23; First posted 2019-07-29 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis C Virus Infection
Keywords: Screening; Telemedicine; Diagnosis
MeSH Terms: conditions — Hepatitis C; Disease

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional care (No Intervention): Screening HCV with dried blod spot (DBS) testing and referral to tertiary care hospital to evaluate disease stage and treatment of HCV RNA positive patients
- Telemedicine care (Active Comparator): Two-way videoconference to evaluate the need of screening with DBS, disease stage evaluation and treatment of HCV RNA positive patients at drug addiction centers
  Interventions: Behavioral: Telemedicine based healthcare programme

INTERVENTIONS:
Behavioral: Telemedicine based healthcare programme — Two-way videoconference to evaluate the need of screening with DBS, disease stage evaluation and treatment of HCV RNA positive patients at drug addiction centers
  Arms: Telemedicine care

SUMMARY:
The investigators have designed a community-based intervention study to all subjects attended in drug addiction centers screened for hepatitis C virus (HCV) to evaluate the efficacy and acceptance of a telemedicine based programme versus conventional healthcare assistance

DETAILED DESCRIPTION:
Our current programme of engagement to healthcare and HCV screening based on on-site dried blood spot (DBS) testing has shown to be successful, but with drop-outs in the HCV cascade of care due to economic reasons that difficulties travel costs to appointments, unconsciousness of disease and low awareness of new direct acting antiviral benefits. In this setting, videoconference as a complement to use of serologic scores and dispensing medication outside the hospital could be useful to improve adherence and reduce drop-outs by reducing the visits to hospital from drug addiction centers (DAC), and promoting direct information regarding benefits of been treated with new antivirals free of interferon directly from specialists.

The hypothesis of the study is that the rate of those diagnosed, fully evaluated of liver disease stage, treated and cured will be improved with a lower rate of drop-outs in the cascade of care in the telemedicine arm compared with the conventional arm without affecting satisfaction in the healthcare assistance process.

This is a prospective, randomized, study in which subjects attending DAC will be invited to participate and sign a consent form.

Aims:

* Evaluation of efficacy (compliance rate with the programme which includes completing screening, liver disease evaluation, and treatment)
* Evaluation of acceptance (grade of patient satisfaction of the programme)
* Evaluation of sustained virological response rate and time to achieve eradication
* The adherence rate to follow-up in participants with advanced fibrosis and cirrhosis
* To assess factors associated with drop-outs
* Cost-effectiveness analysis of the telemedicine programme

Methodology:

The investigators have designed a community-based intervention study to evaluate a telemedicine based programme versus conventional healthcare to all subjects attending DAC and screened for HCV if : a) there is no previous documented HCV antibody request or b) with a previous positive HCV antibody test without viral load (RNA) result or positive result without treatment or confirmed sustained virological response or c) with a negative HCV antibody result tested more than one year ago.

In the conventional arm participants after the dried blood spot (DBS) testing for viral load (RNA) and genotype will be referred to the tertiary care hospital in case of a RNA positive result for a one-day appointment for disease stage evaluation with elastography and prescription of treatment with DBS after12 weeks of finishing treatment for assessing sustained virological response.

In the interventional arm the hepatologist will real-time videoconference with the patient-staff at DAC to discuss the need of DBS for viral load and genotype, evaluation of fibrotic stage by serologic scores and if it is the case in known RNA positive cases prescription of treatment. If DBS is mandatory the patient will be scheduled for a second videoconference to start treatment according to results. Dispensing and custody of treatment will be performed at DAC. Follow-up to assess side effects and sustained virological response will be also scheduled by videoconference.

In both arms when advanced fibrosis or cirrhosis has been detected an appointment at the tertiary care hospital for hepatocellular carcinoma screening will be scheduled every 6 months.

Cost analysis will be performed by investigators to assess medical and non-medical costs and satisfaction of the healthcare model by a validated questionnaire. In all the planned strategies subjects will be asked to complete a questionnaire that includes demographic variables.

For the present study, a 15% improvement in the efficacy (compliance with the programme) was hypothesized in the group of participants receiving the interventional strategy compared to the conventional strategy. Taking into account a power of 80%, alpha error of 5% and losses of 10% will require 83 participants per group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years old or older with a valid sanitary card in our public health system
* Signed Informed consent
* Tested for HCV: a) no previous documented HCV antibody request or b) with a previous positive HCV antibody test without RNA result or positive result without treatment or confirmed sustained virological response or c) with a negative HCV antibody result tested more than one year ago
* No current surveillance by any hepatitis specialized care (hepatology or internal medicine)

Exclusion Criteria:

* Previous DBS testing at DAC lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the intervention | 12 months
  Compliance rate (number of patients of the overall participants) with the programme which includes completing screening, liver disease evaluation, treatment and follow-up visit at 12 week

SECONDARY OUTCOMES:
Acceptance of the intervention with validated satisfaction questionnaire | 12 months
  Grade of patient satisfaction of the telemedicine programme by a validated questionnaire
Sustained virological response rate | 12 months
  Achievement of viral eradication rate (number of patients from the total with active infection that received treatment and achieved eradication)
Time to sustained virological response rate | 12 months
  Time (months) from DBS testing to achievement of viral eradication
Adherence rate to follow-up | 12 months
  Adherence rate (confirmed assistance) to follow-up appointments in patients with advance fibrosis and cirrhosis
Demographic factors associated with drop-outs | 12 months
  Evaluation of demographic characteristics associated with drop-outs in the cascade of care
Cost-effectiveness of telemedicine strategy | 12 months
  Cost-effectiveness analysis taking in consideration utilities and disease management annual costs of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Hernandez-Guerra, MD, Principal Investigator — MD
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Fulgueiras A, Garcia-Pina R, Morant C, de Larrea-Baz NF, Alvarez E. Burden of disease related to hepatitis C and hepatitis B in Spain: a methodological challenge of an unfolding health problem. J Viral Hepat. 2011 Oct;18(10):e453-60. doi: 10.1111/j.1365-2893.2011.01467.x. Epub 2011 Jun 1. PMID 21914063
- [Background] Vallejo F, Barrio G, Brugal MT, Pulido J, Toro C, Sordo L, Espelt A, Bravo MJ; Itinere Project Group. High hepatitis C virus prevalence and incidence in a community cohort of young heroin injectors in a context of extensive harm reduction programmes. J Epidemiol Community Health. 2015 Jun;69(6):599-603. doi: 10.1136/jech-2014-205070. Epub 2015 Apr 13. PMID 25870164
- [Background] Coats JT, Dillon JF. The effect of introducing point-of-care or dried blood spot analysis on the uptake of hepatitis C virus testing in high-risk populations: A systematic review of the literature. Int J Drug Policy. 2015 Nov;26(11):1050-5. doi: 10.1016/j.drugpo.2015.05.001. Epub 2015 Jun 4. PMID 26118799